CLINICAL TRIAL: NCT00121394
Title: Randomized Trial of Chlorhexidine Vaginal and Infant Wash to Reduce Neonatal Mortality
Brief Title: Chlorhexidine Vaginal and Infant Wash in Pakistan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); RTI International (Other); University of Alabama at Birmingham (Other); Aga Khan University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GN 09 A; U01HD040607 (NIH)
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Sepsis; Pregnancy
Keywords: Chlorhexidine; Vaginal wash; Neonatal mortality; Sepsis; Global Network; Maternal and child health; Women's Health; International; Pakistan
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chlorhexidine (Experimental)
  Interventions: Procedure: Chlorhexidine vaginal and infant wash

INTERVENTIONS:
Procedure: Chlorhexidine vaginal and infant wash

SUMMARY:
Infection is a major health problem during birth in Pakistan. This study will look at the possibility of using a septic wash to help improve health during birth in Karachi, Pakistan.

DETAILED DESCRIPTION:
Sepsis in mother and infant is a major cause of perinatal morbidity and mortality in low-resource settings. Several studies have investigated the likelihood that an anti-bacterial agent, chlorhexidine, administered during labor and delivery to mother and infant could reduce the risk of infection and of subsequent maternal and infant morbidity and mortality. In this trial, chlorhexidine wash and placebo will be randomly administered to women in labor and newborn infants in a public hospital in Karachi, Pakistan.

Delivery attendants will administer 0.6% chlorhexidine solution every four hours until delivery (4 washes maximum) and one neonatal wash with the same solution. The control group will receive 200 ml of sterile physiologic saline solution. A total of 5000 women will be randomized in the hospital study, 2500 control and 2500 intervention. All women and infants will be evaluated 24 hours post delivery and at a 7-day follow-up. Women who delivered at home will also receive a 28 days post-partum assessment. Women will be carefully monitored for side effects to the dosage. In addition a community-based feasibility trial of 200 patients (100 CHX, 100 control) will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Gravidas with living fetus delivering at home in the care of identified study birth attendant (community) or admitted to the identified hospital (Civil Hospital Karachi) for delivery

Exclusion Criteria:

* Contraindications to cervical exam (e.g., placenta previa)
* Active genital herpes or vulvovaginal ulceration
* Known or suspected allergy to chlorhexidine
* Fetus with face presentation
* Fetal death
* Unwilling/unable to give informed consent
* Less than 16 years of age

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5008 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Neonatal death or severe sepsis | 7 days

SECONDARY OUTCOMES:
Maternal: clinical chorioamnionitis, clinical endometritis, urinary tract infection, sepsis, length of hospitalization, readmission to hospital, death | 7 days
Neonatal: receipt of antibiotics, duration of hospitalization, readmission to hospital | 7 dats

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldenberg, M.D., Principal Investigator — Drexel University; Sarah Saleem, M.D., Principal Investigator — Aga Khan University
Locations (1):
- Civil Hospital Karachi, Karachi, Pakistan

REFERENCES:
- [Derived] Saleem S, Rouse DJ, McClure EM, Zaidi A, Reza T, Yahya Y, Memon IA, Khan NH, Memon G, Soomro N, Pasha O, Wright LL, Moore J, Goldenberg RL. Chlorhexidine vaginal and infant wipes to reduce perinatal mortality and morbidity: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1225-1232. doi: 10.1097/AOG.0b013e3181e00ff0. PMID 20502294
- [Derived] Saleem S, Reza T, McClure EM, Pasha O, Moss N, Rouse DJ, Bartz J, Goldenberg RL. Chlorhexidine vaginal and neonatal wipes in home births in Pakistan: a randomized controlled trial. Obstet Gynecol. 2007 Nov;110(5):977-85. doi: 10.1097/01.AOG.0000285653.17869.26. PMID 17978107
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org/
- See also: Aga Khan University, Pakistan — http://www.aku.edu/